CLINICAL TRIAL: NCT03462394
Title: Increasing Patient Engagement in the Annual Well Visits Program at NYU Langone Health
Brief Title: Increasing Patient Engagement in the Annual Well Visits Program
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: QI Patient Access Center
Record Dates: First submitted 2018-03-06; First posted 2018-03-12 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Annual Visit, Well Visit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Current Script Version: This arm will receive the version of the call script currently used as part of regular care at NYU Langone Health.
  Interventions: Other: Current Script
- Script Iterations: This arm will receive an iterated version of the script that might contain changes in wording or structure that are different from the current version of the script.
  Interventions: Other: Alternate Script Iterations

INTERVENTIONS:
Other: Current Script — This is the version of the phone call script currently used at NYU Langone Health.
  Groups: Current Script Version
Other: Alternate Script Iterations — Intervention includes various iterations of the phone call script (different wording or script structure).
  Groups: Script Iterations

SUMMARY:
NYU Langone Health calls patients to remind them to schedule their annual well-health appointments (including annual well visit, mammograms, etc.). The proposed study will test different iterations of the call script with the goal of increasing call completion rate and the number of scheduled appointments within an appropriate timeframe.

ELIGIBILITY:
Inclusion Criteria:

* Members attributed to NYU Langone Health under a shared savings arrangement who are due for preventive services and/or screenings and are eligible to be receiving a reminder call.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Members attributed to NYU Langone Health under a shared savings arrangement who are due for preventive services and/or screenings and are eligible to be receiving a reminder call.
Sampling Method: Probability Sample
Enrollment: 5475 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
Number of scheduled annual visits | 6 months

SECONDARY OUTCOMES:
Call completion rate | 6 months
  Call completion rate refers to the percentage of phone calls that successfully complete all steps of the call script.

CONTACTS AND LOCATIONS:
Overall Officials: Leora Horwitz, MD, MHS, Principal Investigator — NYU School of Medicine
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided